CLINICAL TRIAL: NCT02960516
Title: MRI Diffusion Tensor Tractography to Track and Monitor Peripheral Nerve Recovery After Severe Crush or Cut/Repair Nerve Injury
Brief Title: MRI Diffusion Tensor Tractography to Monitor Peripheral Nerve Recovery After Severe Crush or Cut/Repair Nerve Injury
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Wesley Thayer, Wesley Thayer, MD, Phd, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 160761
Record Dates: First submitted 2016-11-06; First posted 2016-11-09 (Estimated); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2022-06

CONDITIONS: Nerve Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MRI of 3.0T — Diffusion Tensor Testing for peripheral nerve monitoring

SUMMARY:
It is estimated that up to 5% of all admissions to level one trauma centers have a peripheral nerve injury. These peripheral nerve injuries may have devastating impacts on quality of life and require months or years to regain function. Neurotmesis, or peripheral nerve transection, is a common injury, with singly cut nerve lacerations accounting for over 60% of the peripheral nerve surgical interventions in civilian studies. For recovery to occur in these patients, axons must grow from the site of repair to the target tissues, a length of up to a meter in humans. By that time, revisional surgery may not be a viable option due to the onset of irreversible muscle atrophy - a transected nerve is estimated to induce a loss of achievable function of approximately 1% for every 6 days of delay. The scenario is even worse for more proximal nerve injuries, such as those that occur in the brachial plexus.

The investigators aim is to longitudinally assess diffusion tensor tractography (DTI) in order to optimize, validate, and translate the ability of DTI to monitor and, more importantly, predict nerve regrowth following trauma and surgical repair. The overall objective of this study is to evaluate the ability of (DTI) to monitor and, more importantly, predict nerve regrowth following crush or cut with surgical repair. The investigators hypothesize that the additional information available via DTI will improve our ability to monitor and predict nerve regrowth following surgical repair or severe crush injury, guiding clinical management either toward or away from surgical intervention.

DETAILED DESCRIPTION:
Although nerve transfers can reduce the length of axonal growth required, failures still occur and revisions are rarely an option due to the aforementioned delays in detection. Current neurodiagnostics [e.g., electromyography (EMG), nerve conduction studies (NCS)] are of limited utility in severely damaged nerves, providing an incomplete picture of nerve microstructural features until target reinnervation occurs. Thus, physicians are limited to a "wait and watch" approach based on qualitative measures obtained from patient history and/or physical exam. This leads to a suboptimal management of peripheral nerve injuries, which in turn can lead to increased instances of irreversible muscle atrophy, paralysis, and/or formation of painful traumatic neuroma.

In terms of the military, extremity injuries accounted for 54% of combat wounds in Operation Iraqi Freedom and Operation Enduring Freedom and recent review of service member injuries during Operation Enduring Freedom noted significant increases in brachial plexus, ulnar, and radial nerve injuries attributable to modern warfare. In addition, symptomatic neuroma occurs in 13% to 32% of amputees, causing pain and limiting or preventing the use of prosthetic devices. Take the example of a wounded warrior with a shrapnel injury to his/her elbow, resulting in the loss of an ulnar nerve segment. Even if nerve grafting is performed, true recovery (motor and/or sensory innervation of the hand) could take up to a year under typical circumstances. If the repair fails, which occurs in up to 40% of patients the failure is typically not truly recognized until that year expires using current management protocols. By that time, revisional surgery is typically not a viable option due to the aforementioned onset of irreversible muscle atrophy. In additional to an inability to effectively monitor nerve recovery after repair, diagnosis of peripheral nerve injuries is difficult using the currently available methods. For example, neurotmesis is a common, but difficult to distinguish, diagnosis following traumatic or iatrogenic extremity injury. Current electrodiagnostic and clinical examinations are invasive, time consuming, and painful. In addition, they cannot perfectly discriminate a severe axonotmetic laceration from a self-resolving neurapraxic injury in the acute setting. This is particularly important in penetrating injuries, or after iatrogenic nerve injuries resulting from nerve blocks, or from intraoperative positioning or external compression, because the degree of axonal injury is unknown.

ELIGIBILITY:
Inclusion Criteria:

subjects between ages of 18 and 64 year of age diagnosed with a Sunderland Class V traumatic neuropathy (transection injury) of the upper extremity nerves that require repair

* Candidates for immediate operative repair of this injury and do not have significant medical comorbidities precluding immediate operative intervention
* willing to comply with all aspects of the treatment (post-operative visits, occupational therapy) and evaluation schedule over the following 12 months
* have peripheral nerve injuries complicated by significant vascular or orthopedic damage

Exclusion Criteria:

* Injuries exhibit gross contamination
* soft tissue coverage is inadequate
* planned staged repair
* have diabetes
* have a neuromuscular disease
* undergoing chemotherapy, radiation therapy or other treatments known to affect the growth of the neural and vascular system
* unlikely to complete occupational therapy
* pregnant or breast-feeding
* subject with any ferromagnetic objects that cannot be removed (cardiac pacemakers, aneurysm clips etc).
* history of claustrophobia

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: subjects between ages of 18 and 64 year of age diagnosed with a Sunderland Class V traumatic neuropathy (transection injury) of the upper extremity nerves that require immediate operative repair of this injury
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Thayer, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Noble J, Munro CA, Prasad VS, Midha R. Analysis of upper and lower extremity peripheral nerve injuries in a population of patients with multiple injuries. J Trauma. 1998 Jul;45(1):116-22. doi: 10.1097/00005373-199807000-00025. PMID 9680023

RESULTS

PARTICIPANT FLOW:
Groups:
- TPNI Group: Subjects who had traumatic peripheral nerve injury (TPNI)
- CTS Group: Participants who had carpal tunnel syndrome (CTS)
- Controls: Healthy control subjects
Period: Overall Study
Arm/Group | TPNI Group | CTS Group | Controls
Started | 3 | 8 | 8
Completed | 3 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TPNI Group | CTS Group | Controls | Total
Number analyzed (Participants) | 3 | 8 | 8 | 19
Age, Customized [Mean (Full Range); unit: years]
  Age | 33.3 [22 to 52] | 53.3 [40 to 73] | 32.4 [20 to 57] | 39.6 [20 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 7 | 13
  Male | 2 | 3 | 1 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Full Range); unit: kg/m^2] | 23.7 [19.7 to 31.8] | 30.5 [23.5 to 38.4] | 25.7 [21 to 32.7] | 26.5 [19.7 to 38.4]

OUTCOME MEASURES:

1. Primary Outcome: Michigan Hand Questionnaire (MHQ) in TPNI Subjects Post Surgery
Description: Michigan Hand Questionnaire assesses hand function and well being of patients with hand injuries.
  It is divided into 6 scales: Overall hand function, scored in a range of 5-25; Activities of daily living, scored in a range of 5-25; Work, scored in a range of 5-25; Pain, scored in a range of 5-25; Aesthetics, scored in a range of 4-16; Satisfaction, scored in a range of 6-30.
  For the pain scale, higher scores indicate more pain. For the other 5 scales, higher scores indicate better hand performance.
  These raw scores are then converted to a range of 0-100 based on the following equations: Overall hand function: -(raw score-25)/20＊100; Activities of daily living: -(raw score-25) 20＊100; Work: (raw score-5)/20＊100; Pain: If question 1=5, then pain score =0; if question 1≠5,then -(raw score-25)/20＊100; Aesthetics:(raw score-4)/16＊100; Satisfaction: -(raw score-30)/24＊100.
  For every patient, an overall MHQ score is obtained by summing the scores for all 6 scales and dividing by 6.
Time Frame: 1, 3, 4, 6, and 9 months post surgery
Population: At each time point only 1 participant was assessed
Measure: Number; unit: score on a scale
Groups:
- Injured Hand in TPNI: Subjects who had traumatic peripheral nerve injury (TPNI), with the assessment being done on the injured hand
- Healthy Hand in TPNI: Subjects who had traumatic peripheral nerve injury (TPNI), with the assessment being done on the healthy (un-injured) hand
Arm/Group | Injured Hand in TPNI | Healthy Hand in TPNI
Number analyzed (Participants) | 1 | 1
score on a scale
  1 month post surgery | 33 | 83
  3 months post surgery | 5 | 75
  4 months post surgery | 69 | 83
  6 months post surgery | 0.8 | 81
  9 months post surgery | 6.8 | 81

2. Primary Outcome: Grip Strength in Subjects With TPNI Post Surgery
Description: The grip strength test is performed by having the participant squeeze as hard as possible on a tool known as dynamometer.
  Grip strength findings were compared between injured and uninjured hands in subjects with TPNI at 3,4, and 6 months post surgery.
  However not all participants were assessed at all time points.
Time Frame: 1, 3, 4, and 6 months post surgery
Population: The overall number of participants was 2; however at each of the time points, only 1 participant was assessed, as presented below.
Measure: Number; unit: pounds
Groups:
- Injured Hand in TPNI: Subjects who had traumatic peripheral nerve injury (TPNI), with the assessment being performed on the injured hand
Arm/Group | Injured Hand in TPNI | Healthy Hand in TPNI
Number analyzed (Participants) | 2 | 2
pounds
  1 month post surgery: number analyzed (Participants) | 1 | 1
  1 month post surgery | NA — Subject was not able to perform test | 92
  3 months post surgery: number analyzed (Participants) | 1 | 1
  3 months post surgery | 30 | 75
  4 months post injury: number analyzed (Participants) | 1 | 1
  4 months post injury | 40 | 100
  6 months post surgery: number analyzed (Participants) | 1 | 1
  6 months post surgery | 18 | 74

3. Primary Outcome: 9 Hole Peg Test in Subjects With TPNI
Description: The Nine Hole Peg Test is used to evaluate patients' fine hand control or dexterity. The total time required to insert nine pegs into nine holes is recorded. The lower the number, the faster the time, the better the performance.
  9HPT findings were compared between injured and uninjured hand at 3,4, and 6 months post surgery in subjects with TPNI. However not all participants were assessed at all time points.
Time Frame: 1, 3, 4, and 6 months post surgery
Population: as for outcome 2
Measure: Number; unit: seconds
Groups:
- Healthy Hand in TPNI: Subjects who had traumatic peripheral nerve injury (TPNI), with the assessment being performed on the healthy (un-injured) hand
Arm/Group | Injured Hand in TPNI | Healthy Hand in TPNI
Number analyzed (Participants) | 2 | 2
seconds
  1 month post surgery: number analyzed (Participants) | 1 | 1
  1 month post surgery | NA — Subject was unable to perform test | 23
  3 months post surgery: number analyzed (Participants) | 1 | 1
  3 months post surgery | 43 | 27
  4 months post surgery: number analyzed (Participants) | 1 | 1
  4 months post surgery | 100 | 27
  6 months post surgery: number analyzed (Participants) | 1 | 1
  6 months post surgery | 51 | 26

4. Primary Outcome: Diffusion Tensor Imaging (DTI) Diffusivity Metrics Post Surgery
Description: Subjects underwent DTI at different time points post surgery; and the metrics analyzed were: Mean Diffusivity (MD), Axial Diffusivity (AD), and Radial Diffusivity (RD).
  Imaging was done to the "healthy" median nerve in controls, injured and healthy (median or ulnar) nerves in patients with TPNI, and compressed median nerve in patients with Carpal Tunnel Syndrome (CTS).
  Imaging was done at multiple timepoints post surgery. Subjects with TPNI underwent imaging at time points falling between 1 and 9 months post surgery. Subjects with CTS underwent imaging at time points falling between 1 and 24 months post surgery. The values were then averaged for each group, as presented below.
Time Frame: Subjects with TPNI underwent imaging at time points falling between 1 and 9 months post surgery. Subjects with CTS underwent imaging at time points falling between 1 and 24 months post surgery.
Measure: Mean (Standard Deviation); unit: μm^2/ms
Groups:
- Injured Nerve-TPNI: Subjects with traumatic peripheral nerve injury, with the imaging being done on the injured nerve
- Healthy Nerve-TPNI: Subjects with traumatic peripheral nerve injury, with the imaging being done on the healthy (un-injured) nerve
- Carpal Tunnel Syndrome (CTS): Subjects diagnosed with carpal tunnel syndrome
- Controls: Healthy subjects who did not have any nerve injury
Arm/Group | Injured Nerve-TPNI | Healthy Nerve-TPNI | Carpal Tunnel Syndrome (CTS) | Controls
Number analyzed (Participants) | 3 | 3 | 8 | 8
μm^2/ms
  Mean Diffusivity (MD) | 1.41 (0.15) | 1.13 (0.28) | 1.27 (0.06) | 1.09 (0.05)
  Axial Diffusivity (AD) | 1.91 (0.19) | 1.82 (0.42) | 1.90 (0.06) | 1.92 (0.05)
  Radial Diffusivity (RD) | 1.16 (0.15) | 0.78 (0.25) | 1.01 (0.06) | 0.67 (0.05)

5. Primary Outcome: Diffusion Tensor Imaging (DTI) Fractional Anisotropy (FA) Metric Post Surgery
Description: Subjects underwent DTI at different time points post surgery and the metric Fractional anisotropy (FA) was analyzed. FA is a scalar value between 0-1 that describe anisotropy of a diffusion process. A value of zero means that diffusion is unrestricted (or equally restricted) in all directions. A value of one means that diffusion occurs only along one axis and is fully restricted along all other directions.
  Imaging was done to the "healthy" median nerve in controls, injured and healthy (median or ulnar) nerves in patients with TPNI, and compressed median nerve in patients with Carpal Tunnel Syndrome (CTS).
  Imaging was done at multiple timepoints post surgery.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Injured Nerve-TPNI | Healthy Nerve-TPNI | Carpal Tunnel Syndrome (CTS) | Controls
Number analyzed (Participants) | 3 | 3 | 8 | 8
score on a scale | 0.32 (0.06) | 0.48 (0.14) | 0.43 (0.03) | 0.59 (0.03)

ADVERSE EVENTS:
Time Frame: Up to 24 months
Arm/Group | TPNI Group | CTS Group | Controls
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/3 | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
We obtained a small cohort, and as such, chose to analyze the data mostly on an individual subject basis. In addition, the affected nerve, injury severity, and treatment varied across TPNI subjects, all of which have a significant impact on outcomes.

The CTS and control groups were not age- and sex-matched, which if done correctly would lead to greater generalizable findings and eliminate the possibility of confounding variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT02960516/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT02960516/ICF_001.pdf